CLINICAL TRIAL: NCT00897546
Title: Multiplex Analysis of Serum Biomarkers for Prediction Interferon Therapy Response in Melanoma Patients
Brief Title: Biomarkers to Predict Response to Interferon Therapy in Patients With Melanoma
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000489213; ECOG-E1L06T1
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma; stage IA melanoma; stage IB melanoma; stage IIA melanoma; stage IIB melanoma; stage IIC melanoma; stage IIIA melanoma; stage IIIB melanoma; stage IIIC melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Collecting and storing samples of blood from patients with cancer to study in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer, and may help doctors learn how well patients will respond to treatment.

PURPOSE: This laboratory study is looking at biomarkers to predict the response to interferon therapy in patients with melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Generate a comprehensive multiplexed array of melanoma-associated serological markers and validate it using serum samples from patients with melanoma and healthy control participants.
* Determine changes in the profile of serological markers induced by interferon-alfa 2b (IFN-α2b) therapy.
* Define panels of serological markers with prognostic and predictive power for IFN-α2b therapy responses in patients with melanoma.

OUTLINE: This is a multicenter study.

Serum samples are used for multiplex analyses. Biomarkers to be assessed include cytokines, chemokines, growth factors, angiogenic and antiangiogenic molecules, matrix metalloproteases (MMPs), tissue inhibitors of MMPs (TIMPs), melanoma-associated antigens, basic fibroblast growth factor, insulin-like growth factor I and II, thrombospondin, endostatin, angiostatin, vasostatin, and vascular endothelial growth factor inhibitor.

PROJECTED ACCRUAL: A total of 1,716 samples will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of melanoma OR healthy volunteer (control)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Samples submitted for research from patients participating in E1690 and E1694
Sampling Method: Non-Probability Sample
Enrollment: 1716 (Actual)
Dates: Start 2007-06-01 (Actual); Primary Completion 2008-07-01 (Actual); Study Completion 2008-07-01 (Actual)

PRIMARY OUTCOMES:
Generation of a comprehensive multiplexed array of melanoma-associated serological markers | 1 month
  Generation of a comprehensive multiplexed array of melanoma-associated serological markers

SECONDARY OUTCOMES:
Changes in the profile of serological markers induced by interferon-alfa 2b therapy | 1 month
  Changes in the profile of serological markers induced by interferon-alfa 2b therapy
Panels of serological markers with prognostic and predictive power for interferon-alfa 2b response | 1 month
  Panels of serological markers with prognostic and predictive power for interferon-alfa 2b response

CONTACTS AND LOCATIONS:
Overall Officials: Elieser Gorelik, MD, PhD, Study Chair — University of Pittsburgh

REFERENCES:
- [Result] Yurkovetsky ZR, Kirkwood JM, Edington HD, Marrangoni AM, Velikokhatnaya L, Winans MT, Gorelik E, Lokshin AE. Multiplex analysis of serum cytokines in melanoma patients treated with interferon-alpha2b. Clin Cancer Res. 2007 Apr 15;13(8):2422-8. doi: 10.1158/1078-0432.CCR-06-1805. PMID 17438101